CLINICAL TRIAL: NCT06939036
Title: A Multicentre, Open-label, Phase I/II Study Investigating the Safety, Tolerability, and Preliminary Efficacy of 225Ac-SSO110 in Participants With Extensive Stage Small Cell Lung Cancer (ES-SCLC) or Merkel Cell Carcinoma (MCC) Receiving Standard of Care (SoC)
Brief Title: Study of 225Ac-SS0110 in Subjects With ES-SCLC or MCC (SANTANA-225 )
Acronym: SANTANA-225
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated due to strategic business decisions.
Sponsor: Ariceum Therapeutics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAX101; 2024-515041-42-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-04

CONDITIONS: Small Cell Lung Cancer Extensive Stage; Merkel Cell Carcinoma
Keywords: actinium; 225Ac; actinium-225; SSO110; SSO120; gallium; 68Ga; gallium-68; radiopharmaceutical; MCC; Merkel Cell carinoma; ES-SCLC; Extensive Stage Small Cell Lung Cancer; radioligand; somatostatin receptor 2; JR11; sstr2-antagonist
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — atezolizumab; durvalumab; avelumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 225Ac-SSO110 + SoC (Experimental)
  Interventions: Drug: 225Ac-SSO110 + SoC; Drug: Atezolizumab; Drug: Durvalumab; Drug: Avelumab; Drug: Pembrolizumab; Drug: Retifanlimab

INTERVENTIONS:
Drug: 225Ac-SSO110 + SoC — Dose Level -2-7
Drug: Atezolizumab — Extensive Stage Small Cell Lung Cancer Checkpoint Inhibitor (SoC)
Drug: Durvalumab — Extensive Stage Small Cell Lung Cancer Checkpoint Inhibitor (SoC)
Drug: Avelumab — Merkel Cell Carcinoma Checkpoint Inhibitor (SoC)
Drug: Pembrolizumab — Merkel Cell Carcinoma Checkpoint Inhibitor (SoC)
Drug: Retifanlimab — Merkel Cell Carcinoma Checkpoint Inhibitor (SoC)

SUMMARY:
This study aims to determine safety, tolerability, recommended phase 2 dose (RP2D), and preliminary antitumor activity of 225Ac-SSO110 with standard of care (SoC) therapy in patients with somatostatin receptor 2 expressing (SSTR2+) extensive-stage small cell lung cancer (ES-SCLC) and recurrent locally advanced or metastatic Merkel cell carcinoma (MCC).

ELIGIBILITY:
Key Inclusion Criteria:

* Signed Informed Consent Form and willing to comply with all study procedures.
* Participants with ES-SCLC (defined as Stage IV per NCCN guidelines Version 1.2024) or recurrent locally advanced or metastatic MCC (per NCCN guidelines Version 1.2024) documented by histology or cytology.
* Participants eligible to receive immune checkpoint inhibitor (CPI) monotherapy at the start of treatment with 225Ac-SSO110 or patients already on CPI monotherapy for 7 weeks.
* ECOG performance status of 0 or 1. Life expectancy of at least 6 months.
* Positive 68Ga-SSO120 scan (Investigator-assessed) during screening.

Key Exclusion Criteria:

* Participants with unstable spinal cord compression.
* Any previous systemic radioligand therapy or extensive radiotherapy.
* Participants receiving or planned to receive consolidative chest radiation.
* History of primary immunodeficiency, transplantation or CAR-T cell therapy.
* Major surgical procedure except diagnostic biopsy within 28 days prior to enrolment or scheduled to have major surgery during the study.
* Inadequate organ or marrow function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Part 1: Safety, tolerability, RP2D of 225Ac-SSO110 in combination with SoC | 42 days
  Identification of the DLT rate per dose level
Part 2: Safety, tolerability, and preliminary anti-tumor activity of 225Ac-SSO110 in combination with SoC at RP2D | 42 days
  Rate of serious adverse events, adverse events, laboratory parameters, and other safety findings, Preliminary anti-tumor activity of 225Ac-SSO110 as assessed by progression free survival (PFS), disease control rate (DCR), best observed response (BOR), overall response rate (ORR), duration of response (DoR)
Part 1 & 2: Safety and tolerability of 68Ga-SSO120 | 7 days
  Rate of serious adverse events, adverse events, laboratory parameters, and other safety findings

CONTACTS AND LOCATIONS:
Locations (7):
- United States (6):
  - Biogenix Molecular, Miami, Florida
  - University of Louisville Health-Brown Cancer Center, Louisville, Kentucky
  - United Theranostics, Glen Burnie, Maryland
  - John Theurer Cancer Center at Hackensack UMC, Hackensack, New Jersey
  - UPMC, Pittsburgh, Pennsylvania
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
- GenesisCare, Alexandria, Australia

IPD SHARING:
Plan to Share IPD: Yes